CLINICAL TRIAL: NCT03183076
Title: Efficacy, Tolerability and Adherence of the Modified Atkins Diet on Drug-resistant Epilepsy in Adults Patients
Brief Title: Efficacy, Tolerability and Adherence of the Modified Atkins Diet on Drug-resistant Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, María Ingrid Alanis Guevara, MD neurologist, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: F2016-1301-72
Record Dates: First submitted 2017-05-31; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Epilepsy, Drug Resistant
Keywords: epilepsy; Diet, Carbohydrate-Restricted; Drug Resistance
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy | interventions — Drug Therapy; Diet; Therapeutics; Anticonvulsants

STUDY DESIGN:
Intervention Model Description: Clinical trial, Parallel, controled
Who Masked: Investigator
Masking Description: MD María Ingrid Alanis Guevara. Neurologist Hospital of the Western National Medical Center. Guadalajara. Mexico
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified adkins diet (Active Comparator): modified adkins diet. It consists in the free intake of proteins and fats, and the restriction of carbohydrates that are gradually being installed. Its mechanism of action that induces a state of ketosis.
  Interventions: Other: modified adkins diet
- Pharmacotherapy without diet (Active Comparator): It consists in administer only pharmacological treatment withot a special diet, Drug-resistant epilepsy is characterized by the use of antiepileptic drugs and in optimal doses, depending on the type of epilepsy, at least on two consecutive occasions without response to management.
  Interventions: Drug: Pharmacotherapy without diet

INTERVENTIONS:
Other: modified adkins diet — Patients were assigned to two groups, one of them received modified adkins diet for treatment of drug-resistant epilepsy. It consists in the free intake of proteins and fats, and the restriction of carbohydrates that are gradually being installed. Its mechanism of action that induces a state of ketosis
  Other Names: adkins diet in drug-resistant epilepsy
  Arms: modified adkins diet
Drug: Pharmacotherapy without diet — Patients were assigned to two groups, one of them received conventional treatment with antiepileptic drugs without a special diet
  Other Names: treatment with antiepileptic drugs
  Arms: Pharmacotherapy without diet

SUMMARY:
The Atkins Diet Modified (ADM) is the best alternative treatment for drug-resistant epilepsy, There is a high prevalence worldwide , especially in Latin American countries, including Mexico.

Low income earners, many of which do not have a social security, must meet the high costs by Antiepileptic Drugs (AEDS), which in addition should be used in conjunction or combination therapy, because monotherapy is insufficient .

The diet adkins makes some changes in the traditional food habits by others that are accessible and not necessarily expensive, whose mechanism allows for better control of the seizures.

DETAILED DESCRIPTION:
Objective: To assess the efficacy, tolerability and adherence of the modified adkins diet in adult patients with drug-resistent epilepsy Materials and Methods: Clinical trial, made up of patients with drug-resistent epilepsy, selected by convenience, who will be handled pharmacologically with the standard treatment of this condition for a period of not less than 6 months, after which they will be treated with adkins diet modified, prior informed consent, to establish its effect and a comparative analysis later.

The objective of this work is to analyze the efficacy, tolerability and adherence of the modified atkins diet in adult patients with drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Patients that meet the criteria of drug-resistant epilepsy
* Patients treated with Rational polytherapy, a minimum of 6 months, with no changes in their drug refractory condition.
* Patients with drug- resistant epilepsy with informed consent signed by themselves and their proxy.
* Patients with drug-resistant epilepsy of any etiology, except tumor, metabolic, degenerative or progressive.

Exclusion Criteria:

* Patients with drug-resistant epilepsy simultaneous alternate treatment to the Atkins Diet modified.
* Patients with a neurological entity progressive and fatal
* Patients with congenital diseases and difficulty to metabolize fats or that require high amounts of carbohydrates in the diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Frequency of epileptic seizures | 3 months
  Frequency of epileptic seizures measured according to the clinical criteria of therapeutic evaluation of Huttenlocher

SECONDARY OUTCOMES:
Therapeutic response observed in electroencephalogram | 3 months
  Panic electroencephalographic criteria on the therapeutic response. Having regard to the standardization, improvement or worsening of the crisis in the electroencephalogram
Measurement of quality of life and decrease in seizures | 3 months
  Interrogate the patient with a questionnaire of refractory epilepsy drugs. And ask to the patient with this questionnaire if improved their quality of life and have decreased seizures after using the atkins diet modified.
Blood tests (Hematic biometry) | 3 months
  Take this blood test to assess the general conditions of the patient and see their levels of hemoglobin, hematocrit, leukocyte and platelet count.
Blood chemistry (serum electrolytes) | 3 months
  It will evaluate the general condition of the patient and with this test rule out the presence of electrolyte imbalance
liver function tests | 3 months
  Will be evaluated with this test levels of transaminases as can be raised by treatment anticonvulsant and see if there are any changes with the changes in the diet of patients
ketonuria | 3 months
  It will assess the levels of ketones in urine due to the change in the diet of patients with the Atkins diet

CONTACTS AND LOCATIONS:
Overall Officials: María I Alanis, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Western Medical Center, Mexican Institute of Social Security, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Proposal for revised classification of epilepsies and epileptic syndromes. Commission on Classification and Terminology of the International League Against Epilepsy. Epilepsia. 1989 Jul-Aug;30(4):389-99. doi: 10.1111/j.1528-1157.1989.tb05316.x. No abstract available. PMID 2502382
- [Background] Panico LR, Rios VG, Demartini MG, Carniello MA. [The electroencephalographic evolution of a group of patients on a ketonic diet]. Rev Neurol. 2000 Jan 1-15;30(1):8-15. Spanish. PMID 10742989
- [Background] Freeman J, Veggiotti P, Lanzi G, Tagliabue A, Perucca E; Institute of Neurology IRCCS C. Mondino Foundation. The ketogenic diet: from molecular mechanisms to clinical effects. Epilepsy Res. 2006 Feb;68(2):145-80. doi: 10.1016/j.eplepsyres.2005.10.003. PMID 16523530
- [Background] Kossoff EH, Zupec-Kania BA, Amark PE, Ballaban-Gil KR, Christina Bergqvist AG, Blackford R, Buchhalter JR, Caraballo RH, Helen Cross J, Dahlin MG, Donner EJ, Klepper J, Jehle RS, Kim HD, Christiana Liu YM, Nation J, Nordli DR Jr, Pfeifer HH, Rho JM, Stafstrom CE, Thiele EA, Turner Z, Wirrell EC, Wheless JW, Veggiotti P, Vining EP; Charlie Foundation, Practice Committee of the Child Neurology Society; Practice Committee of the Child Neurology Society; International Ketogenic Diet Study Group. Optimal clinical management of children receiving the ketogenic diet: recommendations of the International Ketogenic Diet Study Group. Epilepsia. 2009 Feb;50(2):304-17. doi: 10.1111/j.1528-1167.2008.01765.x. Epub 2008 Sep 23. PMID 18823325
- [Result] Berg AT, Kelly MM. Defining intractability: comparisons among published definitions. Epilepsia. 2006 Feb;47(2):431-6. doi: 10.1111/j.1528-1167.2006.00440.x. PMID 16499772
- [Result] Brodie MJ, Kwan P. Staged approach to epilepsy management. Neurology. 2002 Apr 23;58(8 Suppl 5):S2-8. doi: 10.1212/wnl.58.8_suppl_5.s2. PMID 11971127
- [Result] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Result] Kwan P, Brodie MJ. Definition of refractory epilepsy: defining the indefinable? Lancet Neurol. 2010 Jan;9(1):27-9. doi: 10.1016/S1474-4422(09)70304-7. Epub 2009 Nov 13. No abstract available. PMID 19914135
- [Result] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Result] Martinez-Juarez IE, Lopez-Zapata R, Gomez-Arias B, Bravo-Armenta E, Romero-Ocampo L, Estevez-Cruz Z, Hernandez-De la Cruz G, Moran-Molina S. [Refractory epilepsy: use of the new definition and related risk factors. A study in the Mexican population of a third-level centre]. Rev Neurol. 2012 Feb 1;54(3):159-66. Spanish. PMID 22278892
- [Result] Shorvon SD. The epidemiology and treatment of chronic and refractory epilepsy. Epilepsia. 1996;37 Suppl 2:S1-S3. doi: 10.1111/j.1528-1157.1996.tb06027.x. PMID 8641240
- [Result] Devinsky O. Patients with refractory seizures. N Engl J Med. 1999 May 20;340(20):1565-70. doi: 10.1056/NEJM199905203402008. No abstract available. PMID 10332020
- [Result] Arroyo S. [Evaluation of drug-resistant epilepsy]. Rev Neurol. 2000 May 1-15;30(9):881-6. Spanish. PMID 10870204
- [Result] Benbadis SR, Tatum WO, Vale FL. When drugs don't work: an algorithmic approach to medically intractable epilepsy. Neurology. 2000 Dec 26;55(12):1780-4. doi: 10.1212/wnl.55.12.1780. No abstract available. PMID 11188984
- [Result] Hauser WA. The natural history of drug resistant epilepsy: epidemiologic considerations. Epilepsy Res Suppl. 1992;5:25-8. PMID 1418457
- [Result] Marson AG, Appleton R, Baker GA, Chadwick DW, Doughty J, Eaton B, Gamble C, Jacoby A, Shackley P, Smith DF, Tudur-Smith C, Vanoli A, Williamson PR. A randomised controlled trial examining the longer-term outcomes of standard versus new antiepileptic drugs. The SANAD trial. Health Technol Assess. 2007 Oct;11(37):iii-iv, ix-x, 1-134. doi: 10.3310/hta11370. PMID 17903391
- [Result] Sanchez-Alvarez JC, Serrano-Castro P, Canadillas-Hidalgo F. [Refractory epilepsy in adults]. Rev Neurol. 2002 Nov 16-30;35(10):931-53. Spanish. PMID 12436398
- [Result] Serrano Castro PJ, Sanchez Alvarez JC. [Controversies about the new anti-epileptic drugs]. Rev Neurol. 2001 Jan 16-31;32(2):165-71. Spanish. PMID 11299481
- [Result] Gomez-Alonso J, Giraldez BG. [Epilepsy: a new definition for an old disease]. Rev Neurol. 2007 Jul 16-31;45(2):126-7. No abstract available. Spanish. PMID 17642053
- [Result] Fisher RS, van Emde Boas W, Blume W, Elger C, Genton P, Lee P, Engel J Jr. Epileptic seizures and epilepsy: definitions proposed by the International League Against Epilepsy (ILAE) and the International Bureau for Epilepsy (IBE). Epilepsia. 2005 Apr;46(4):470-2. doi: 10.1111/j.0013-9580.2005.66104.x. PMID 15816939
- [Result] Hefft S, Jonas P. Asynchronous GABA release generates long-lasting inhibition at a hippocampal interneuron-principal neuron synapse. Nat Neurosci. 2005 Oct;8(10):1319-28. doi: 10.1038/nn1542. Epub 2005 Sep 11. PMID 16158066
- [Result] Hestrin S, Galarreta M. Synchronous versus asynchronous transmitter release: a tale of two types of inhibitory neurons. Nat Neurosci. 2005 Oct;8(10):1283-4. doi: 10.1038/nn1005-1283. No abstract available. PMID 16189532
- [Result] Callaghan BC, Anand K, Hesdorffer D, Hauser WA, French JA. Likelihood of seizure remission in an adult population with refractory epilepsy. Ann Neurol. 2007 Oct;62(4):382-9. doi: 10.1002/ana.21166. PMID 17880009
- [Result] Duncan JS. The outcome of epilepsy surgery. J Neurol Neurosurg Psychiatry. 2001 Apr;70(4):432. doi: 10.1136/jnnp.70.4.432. No abstract available. PMID 11254763
- [Result] Huttenlocher PR, Wilbourn AJ, Signore JM. Medium-chain triglycerides as a therapy for intractable childhood epilepsy. Neurology. 1971 Nov;21(11):1097-103. doi: 10.1212/wnl.21.11.1097. No abstract available. PMID 5166216
- [Result] Panico LR, Demartini MG, Rios VG, Carniello MA. [The ketogenic diet in infantile refractory epilepsy: electroclinical response, complications and secondary effects]. Rev Neurol. 2000 Aug 1-15;31(3):212-20. Spanish. PMID 10996924
- [Result] Lefevre F, Aronson N. Ketogenic diet for the treatment of refractory epilepsy in children: A systematic review of efficacy. Pediatrics. 2000 Apr;105(4):E46. doi: 10.1542/peds.105.4.e46. PMID 10742367
- [Result] Vicente-Hernandez M, Garcia-Garcia P, Gil-Nagel A, Lopez-Munoz F, Alamo C. [Therapeutic approach to epilepsy from the nutritional view: current status of dietary treatment]. Neurologia. 2007 Oct;22(8):517-25. Spanish. PMID 17641989
- [Result] Yudkoff M, Daikhin Y, Melo TM, Nissim I, Sonnewald U, Nissim I. The ketogenic diet and brain metabolism of amino acids: relationship to the anticonvulsant effect. Annu Rev Nutr. 2007;27:415-30. doi: 10.1146/annurev.nutr.27.061406.093722. PMID 17444813
- [Derived] Martin-McGill KJ, Bresnahan R, Levy RG, Cooper PN. Ketogenic diets for drug-resistant epilepsy. Cochrane Database Syst Rev. 2020 Jun 24;6(6):CD001903. doi: 10.1002/14651858.CD001903.pub5. PMID 32588435